CLINICAL TRIAL: NCT02791997
Title: Consequences of a Brain Lesion or of Migraine on Auditory Processing: Attention, Memory and Emotion
Brief Title: Audition After a Lesion and in Migraine. (AuditionPostLesion)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL14_0202; 2014-A01289-38 (Other: ID-RCB)
Record Dates: First submitted 2016-05-27; First posted 2016-06-07 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2022-08

CONDITIONS: Migraine Disorders, Brain
Keywords: Audition; Stroke; Migraine; Attention; Short-term memory,; Emotions; EEG; MEG
MeSH Terms: conditions — Migraine Disorders; Stroke | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brain-damaged patients (Experimental)
  Interventions: Other: Neuropsychological tests; Other: Neurophysiological tests
- Control participants (Experimental)
  Interventions: Other: Neuropsychological tests; Other: Neurophysiological tests
- Migraine patients (Experimental)
  Interventions: Other: Neuropsychological tests; Other: Neurophysiological tests

INTERVENTIONS:
Other: Neuropsychological tests — Neuropsychological tests consist in listening to sounds in various contexts and providing behavioral responses with response-buttons.
Other: Neurophysiological tests — Neurophysiological tests consist in the recording of EEG and/or MEG signals while realizing the neuropsychological tests, as well as MRI scanning to characterize the patients' brain lesions and reconstruct the brain sources of surface EEG/MEG signals.

SUMMARY:
The project studies auditory processing after brain damage (in temporal and/or frontal areas) and in migraine. The auditory processes investigated are attention, short-term memory, sound-induced emotions. To characterize auditory deficits after brain damage or in migraine, neuropsychological assessments are combined with neurophysiological markers (Electro-encephalography: EEG, Magneto-encephalography: MEG, Magnetic Resonance Imaging: MRI).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 80
* MEG/MRI compatibility
* Motivation to participate efficiently in the study
* No severe hearing loss
* Informed consent to participate in the study
* Affiliation to social security
* For brain-damaged patients : no need for medical assistance; focal temporal and/or frontal lesion; no major cognitive impairment; ability to understand and apply the instructions for neuropsychological testing; testing at least one-month after the event resulting in brain damage; absence of neurological and psychiatric disorders besides the lesion
* For migraine patients: no need for medical assistance; migraine diagnosis; no major cognitive impairment; ability to understand and apply the instructions for neuropsychological testing; absence of neurological and psychiatric disorders besides the migraine
* Healthy participants: absence of neurological and psychiatric disorders

Exclusion Criteria:

* Age below 18 or above 80
* MRI scanning not possible: artificial cardiac pacemaker, insulin pump, metallic prosthesis, intra-cerebral clip, claustrophobia
* MEG acquisition not possible: large heads, neurostimulator, metal in the head or the body.
* Pregnant or breast-feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Percentages of correct responses in Neuropsychological tests | up to 2 months
reaction times in Neuropsychological tests | up to 2 months

SECONDARY OUTCOMES:
Event-Related Potentials (EEG) in Neurophysiological tests | up to 2 months
Event-Related Fields (MEG) in Neurophysiological tests | up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Norbert NIGHOGHOSSIAN, MD, Principal Investigator — Unité 201, Hôpital Neurologique, Hospices Civils de Lyon
Locations (2):
- France (2):
  - Unité 201, Hôpital Neurologique, Bron
  - Service Explorations Fonctionnelles Neurologiques, Hôpital de la Croix-Rousse, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Masson R, Demarquay G, Meunier D, Leveque Y, Hannoun S, Bidet-Caulet A, Caclin A. Is Migraine Associated to Brain Anatomical Alterations? New Data and Coordinate-Based Meta-analysis. Brain Topogr. 2021 May;34(3):384-401. doi: 10.1007/s10548-021-00824-6. Epub 2021 Feb 19. PMID 33606142